CLINICAL TRIAL: NCT02598609
Title: Study on Preventing Adverse Events in Neonates (SEPREVEN): a Stepped-wedge Randomised Controlled Trial to Reduce Adverse Event Rates in the NICU
Brief Title: SEPREVEN: a Stepped-wedge Randomised Controlled Trial
Acronym: SEPREVEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Caeymaex Laurence (Other)
Collaborators: Paris 12 Val de Marne University (Other); Ministry of Health, France (Other Government)
Responsible Party: Sponsor-Investigator, Dr Caeymaex Laurence, Dr, PhD, Centre Hospitalier Intercommunal Creteil
Organization: Centre Hospitalier Intercommunal Creteil (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SEPREVEN
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Intensive Care Units, Neonatal; Misadventures to Patients During Surgical and Medical Care; Catheter-related Bloodstream Infection (CRBSI) Nos; Quality of Healthcare; Ventilator Adverse Event; Nosocomial Pneumonia; Immature Newborn; Skin Lesion; Extravasation Injury; Nasal Injury; Intubation Complication; Medication Administered in Error; IV Catheter Nos Deep Venous Thrombosis
Keywords: Adverse event; Neonatal Intensive Care Unit; Catheter-related Bloodstream Infection (CRBSI) nos; Extravasation injury; Medication error; Central venous catheter complication; Unprogrammed extubation
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Healthcare-Associated Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cluster A (Other): Out of the 12 participating NICUs, 4 NICUs are randomly assigned in Cluster A. The intervention (educational program for preventing adverse events and medical errors in the NICU) is implemented after a pre interventional period of 4 months. The intervention is implemented during 4 months. The length of the post interventional period is 12 months.
  Interventions: Behavioral: Education program for NICU caregivers
- Cluster B (Other): Out of the 12 participating NICUs, 4 NICUs are randomly assigned in Cluster B. The intervention (educational program for preventing adverse events and medical errors in the NICU) is implemented after a pre interventional period of 8 months. The intervention is implemented during 4 months. The length of the post interventional period is 8 months.
  Interventions: Behavioral: Education program for NICU caregivers
- Cluster C (Other): Out of the 12 participating NICUs, 4 NICUs are randomly assigned in Cluster C. The intervention (educational program for preventing adverse events and medical errors in the NICU) is implemented after a pre interventional period of 12 months. The intervention is implemented during 4 months. The length of the post interventional period is 4 months.
  Interventions: Behavioral: Education program for NICU caregivers

INTERVENTIONS:
Behavioral: Education program for NICU caregivers — * standardized educational program : learning how to retrospectively analyze causes of a medical error in the NICU in order to prevent it (compulsory)
  * implementation of a central line maintenance bundle and checklist, of a central line insertion bundle and checklist and of a daily goals bundle and checklist. (compulsory)
  * poster for prevention of extravasation injuries

SUMMARY:
Adverse events are frequent in Neonatal Intensive Care Units' (NICU) patients and account for a high morbidity and mortality. Possible severe adverse events are central line associated bloodstream infections (CLABSI), ventilator and catheter associated adverse events and medication errors. Severity of the patient's outcome after an adverse event can be classified using the National Coordinating Council for Medication Error Reporting and Preventing (NCC MERP) Index for categorizing medication errors.

The study will test the hypothesis that rates of adverse events in NICU patients will be reduced by the implementation of an educational program for the NICU caregivers (nurses and physicians), consisting of strategies for recognizing and preventing adverse events in their unit. These strategies will be oriented to prevent CLABSI, medication errors, skin and nasal complications and ventilator and catheter-associated adverse events.

This trial has a stepped wedge cluster design, in which the NICUs from 12 hospitals in France will be randomized to the timing of implementation of the educational program.

In order to describe the adverse events occurring during the study period, an anonymous voluntary adverse event reporting system will be provided to the caregivers of the participating units. A nested study will examine how caregivers communicate with the patients' parents in case of adverse event (disclosure or not, and caregivers' reasons).

The rates of adverse events will be measured retrospectively using a neonatal NICU trigger tool.

ELIGIBILITY:
Inclusion Criteria :

* Patients hospitalized during the study period in one of the 12 participating Neonatal Intensive Care Units
* Corrected Gestational age not exceeding 42 weeks +6 days at the time of admission in the NICU
* Length of hospitalisation in the NICU > 2 days
* No parental objection to the anonymous data collection of their newborn(s)' clinical data, after written information

Exclusion Criteria:

* More than 42 weeks +6 days of corrected gestational age on admission in the NICU
* Length of hospitalization in the NICU < or = 2 days
* Parental objection to the anonymous data collection of their newborn(s)' clinical data

Ages: 1 Day to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8000 (Estimated)
Dates: Start 2015-11-23 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Rates of adverse events (total number/1000 patient-days) | 20 months
  Assessment of the effectiveness of the program on reducing the rates of adverse events (number of adverse events/1000 patient-days) (AEs) measured using a retrospective chart review with a NICU trigger tool (Sharek PJ et al. Pediatrics 2006;118(4):1332-1340). Out of the pool of patients included in the study, 3600 charts (60 charts per 4 months and per unit) will be randomly assigned to be reviewed using the NICU trigger tool. An adverse event is defined here as an injury, large or small, caused by the use (including non-use) of a drug, test, or medical treatment.(Trigger tool kit, Raju Ped Research). Preventable adverse events and non preventable adverse events secondary to expected complications or side effects are both included.

SECONDARY OUTCOMES:
Rate of adverse events (Percentage of patient admissions with an adverse event) over time during the study period | 20 months
  Assessment of the effectiveness of the program on reducing the rate of adverse events (percentage of patient admissions with an adverse event) measured using a retrospective chart review with a NICU trigger tool (Sharek PJ et al. Pediatrics 2006;118(4):1332-1340), over time during the inclusion period
Rate of adverse events (number of adverse events per 100 NICU admissions) over time during the study period | 20 months
  Assessment of the effectiveness of the program on reducing the rates of adverse events (number of adverse events per 100 admissions) (AEs) measured using a retrospective chart review with a NICU trigger tool (Sharek PJ et al. Pediatrics 2006;118(4):1332-1340) over time
Rates of preventable adverse events (total number/1000 patient-days) | 20 months
  Assessment of the effectiveness of the program on reducing the rates of preventable adverse events (number of adverse events/1000 patient-days) (AEs) measured using a retrospective chart review with a NICU trigger tool (Sharek PJ et al. Pediatrics 2006;118(4):1332-1340). Out of the pool of patients included in the study, 3600 charts (60 charts per 4 months and per unit) will be randomly assigned to be reviewed using the NICU trigger tool. An adverse event is defined here as an injury, large or small, caused by the use (including non-use) of a drug, test, or medical treatment. (see Trigger tool kit definitions and Raju Ped Research) Preventability is assessed according to the existence of an "error". Expected complications or side effects from therapeutic or diagnostic interventions are generally non-preventable, and hence are considered complications. (see Raju, Pediatric Research) Healthcare associated infections are considered preventable adverse events.
Rates of CLABSI, number per 1000 catheter-days in the 12 participating NICUs in France | 20 months
  Assessment of the effectiveness of the program on reducing the rates of Central line associated blood stream infections defined using the Primary Blood Stream Infections and LCBSI criteria (CDC/NHSN Device-Associated Module BSI January 2015), collected prospectively in the 12 participating NICUs. Analysis will include subgroups according to patient's characteristics and contextual factors (nurse staffing, unit occupancy, type of unit).
Rates of unplanned extubations, number per 100 ventilator-days and number per 100 ventilator-hours in the 12 participating NICUs in France. | 20 months
  Assessment of the effectiveness of the program on reducing the rates of adverse events caused/lead by unplanned extubations measured using the retrospective trigger tool chart review (Sharek PJ et al. Pediatrics 2006;118(4):1332-1340). Out of the pool of patients included in the study, 3600 charts (60 charts per 4 months and per unit) will be randomly assigned to be reviewed using the NICU trigger tool.
Identify factors associated with and consequences of Unprogrammed extubation in NICU patients | 20 months
  Unprogrammed extubation: description of prospectively reported factors associated with UE (context and cause), and patients' characteristics, as well as HCP's assessment of preventability of this UE (multiple choices questionnaire) in the participating units. Prospective collection of outcome 30 minutes and 24 hours after UE (reintubation/ non invasive ventilation or spontaneous breathing and outcome severity grading) according to reported causal factors and patients' characteristics
Rates of severe adverse events | 20 months
  Assessment of the effectiveness of the program on reducing the rates of severe adverse events collected using a multisource prospective voluntary anonymous collection. Results will include control charts, and include patients' characteristics and contextual factors over time.
Describe rates of medication errors in NICU patients | 20 months
  Assessment of the effectiveness of the program on reducing the rates of adverse events related to medication errors, measured using the retrospective trigger tool chart review (Sharek PJ et al. Pediatrics 2006;118(4):1332-1340). Out of the pool of patients included in the study, 3600 charts (60 charts per 4 months and per unit) will be randomly assigned to be reviewed using the NICU trigger tool; A medication error is defined here as any preventable event that causes or leads to inappropriate medication use with patient harm while the medication is in the control of the health care professional in the NICU. (see Raju Ped Research).
Identify factors associated with and consequences of medication errors in NICU patients | 20 months
  Type of medication, of error and consequences and patients' and unit's characteristics are collected prospectively in the participating NICUs
Identify factors associated with and consequences of catheter-related adverse in the NICU | 20 months
  Type of adverse event, consequence and patients' and unit's characteristics are collected prospectively in the participating NICUs
Rates of catheter-related adverse events, number per 1000 catheter-days | 20 months
  Assessment of the effectiveness of the program on reducing the rates of catheter-related adverse events collected prospectively and using the retrospective trigger tool chart review (Sharek PJ et al. Pediatrics 2006;118(4):1332-1340) in the 12 participating NICUs
Identify number and types of medical errors collected in the 12 NICUs in France | 20 months
  Number and types of medical errors are defined as catheter related (central line), medication, ventilation, skin lesions, nasal injury, extravasation, enteral feeding, temperature control, unprogrammed extubation, surgical complications, diagnostic error or delay, parenteral fluid/nutrition adverse event, and, in existing, others. These "errors" are collected prospectively in each participating unit during the 20 months period, using a multi-source collection file (manual, anonymous and voluntary and/or institutional). A Medical Error is defined here as an error in health care, due to a failure of the planned action to be completed as intended, or using a wrong plan of action to achieve the goal, and excluding near misses. (see Raju Pediatric Research) Errors are included independently of the harm caused to the patient. Descriptions will include patients' characteristics and contextual factors.
Identify Severity of adverse events in the 12 participating NICUs in France | 20 months
  Identify Severity of adverse events, rated prospectively using the National Coordinating Council for Medication Error Reporting and Prevention Index for Categorizing Errors (NCC MERP, 2001)(including infectious and non infectious adverse events). Severity is described according to contextual factors and patients' characteristics.
Describe late-onset infections types and characteristics in NICU patients in France | 20 months
  Late-onset infections are defined according to the January 2015 CDC/NHSN Surveillance Definitions for all types of Specific Types of infections, for Primary Blood Stream Infections and for neonatal Ventilator associated pneumonia (Hospital-Acquired infections for neonates). Clinical sepsis without laboratory proven infection is included. Description includes type on infection, clinical and bacteriological characteristics and type of consequence - data are collected prospectively by physicians. Descriptions will be done including patients' characteristics and contextual factors.
Skin tolerance to cutaneous antisepsis : Dermatitis score results before and after an antisepsis procedure for umbilical and/or PICC catheter insertion in premature neonates born less than 32 weeks gestational age and aged less than 15 days. | 20 months
  Dermatitis scoring is based on the existing Dermatitis score used by Garland JS (Garland JS et al. J Perinatol 2009), traduced in french (Score sheet available on demand). Score ranges from 0 (no dermatitis) to 4, with severe dermatitis >= 2. Score is completed propectively by the nurse in care, before and untill 5 after the procedure. Scores wil be compared according to antiseptic procedure and patient's characteristics.
Description of Nasal scores results during the use of noninvasive nasal ventilation interfaces in neonates born less than 32 weeks of gestational age and aged less than 15 days | 20 months
  The nasal trauma score is based on the score used by Collins (Collins CL et al, Eur J Ped 2014). Score is completed prospectively by the nurse in care of the patient, in the first week of nasal ventilation (after extubation or not). Rates and type of nasal lesions according to interface and patient's characteristics will be described.
Identify characteristics ad factors associated with severe extravasation injuries in the 12 NICUs | 20 months
  Extravasation injuries from peripherally inserted short catheter score is rated from I to IV based on the classification described b are collected prospectively using the score described by Casanova (Casanova D et al, Br J Plastic Surgery 2001). Score is rated prospectively by nurse in care; for severe extravasation, context of extravasation (infused substances, site,...), patients' characteristics and consequences are collected prospectively.
Description of characteristics of disclosed and undisclosed adverse events to the patients' parents, caregivers' motivations, and perceived parental reactions | 20 months
  For each collected adverse event, caregivers self-administered written questionnaire assessing of adverse event has been told to parent(s), heath care professional's reasons to disclosure it or not, and in case of disclosure, parental reactions according to health care professional (multiple choices)
Economical impact of the program | 20 months
  Mortality (yes/no)
Economical impact of the program | 20 months
  NICU length of stay (days)
Economical impact of the program | 20 months
  Neurological complications (Intraventricular hemorrhage, leucomalacia) for prematures
Economical impact of the program | 20 months
  Hospitalization data: morbidity for prematures bronchopulmonary dysplasia at 36 weeks (yes/no); severe retinopathia (yes/no); severe enterocolitis (yes/no)
Rate of positive and negative blood cultures in NICU patients suspected of late onset infection according to volume of blood culture | 20 months
  Prospective record on volume of blood culture and results (positive/negative)
Description of safety culture in each of the 12 participating NICUs before and after patients' inclusion period | 20 months
  Safety culture is measured by a questionnaire filled in by the healthcare providers of the 12 units, in the weeks before the beginning and after the end of the patients' inclusion period using the french traduction of the Hospital Survey On Patient Safety Culture (HSOPSC)(http://www.ahrq.gov/qual/patientsafetyculture), named Questionnaire de mesure de la culture de sécurité des soins en milieu hospitalier, validated by the CCECQA. A comparison of the results before and after the study will be described globally and per unit.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Caeymaex, MD, PhD, Principal Investigator — CHI Creteil, Paris Est University
Locations (12):
- France (12):
  - CHU Strasbourg Hautepierre, Strasbourg, Alsace
  - CHU Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - CHU Lille Jeanne de Flandres, Lille, Hauts-de-France
  - CHU Caen, Caen, Normandy
  - CHU Angers, Angers, Pays de la Loire Region
  - CHU Nice Archet, Nice, Provence-Alpes-Côte d'Azur Region
  - CHI Creteil, Créteil, Île-de-France Region
  - CHU Bicêtre, APHP, Le Kremlin-Bicêtre, Île-de-France Region
  - CHU Robert Debré, APHP, Paris, Île-de-France Region
  - CH Poissy, Poissy, Île-de-France Region
  - CH Pontoise René Dubos, Pontoise, Île-de-France Region
  - Centre Hospitalier Delafontaine, Saint-Denis, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharek PJ, Horbar JD, Mason W, Bisarya H, Thurm CW, Suresh G, Gray JE, Edwards WH, Goldmann D, Classen D. Adverse events in the neonatal intensive care unit: development, testing, and findings of an NICU-focused trigger tool to identify harm in North American NICUs. Pediatrics. 2006 Oct;118(4):1332-40. doi: 10.1542/peds.2006-0565. PMID 17015521
- [Background] Sharek PJ. The Emergence of the Trigger Tool as the Premier Measurement Strategy for Patient Safety. AHRQ WebM&M. 2012 May 1;2012(5):120. No abstract available. PMID 23667349
- [Background] Chedoe I, Molendijk H, Hospes W, Van den Heuvel ER, Taxis K. The effect of a multifaceted educational intervention on medication preparation and administration errors in neonatal intensive care. Arch Dis Child Fetal Neonatal Ed. 2012 Nov;97(6):F449-55. doi: 10.1136/fetalneonatal-2011-300989. Epub 2012 Apr 5. PMID 22491014
- [Background] Dabliz R, Levine S. Medication safety in neonates. Am J Perinatol. 2012 Jan;29(1):49-56. doi: 10.1055/s-0031-1285831. Epub 2011 Aug 22. PMID 21861251
- [Background] Palmero D, Di Paolo ER, Beauport L, Pannatier A, Tolsa JF. A bundle with a preformatted medical order sheet and an introductory course to reduce prescription errors in neonates. Eur J Pediatr. 2016 Jan;175(1):113-9. doi: 10.1007/s00431-015-2607-4. Epub 2015 Aug 15. PMID 26272253
- [Background] Fisher D, Cochran KM, Provost LP, Patterson J, Bristol T, Metzguer K, Smith B, Testoni D, McCaffrey MJ. Reducing central line-associated bloodstream infections in North Carolina NICUs. Pediatrics. 2013 Dec;132(6):e1664-71. doi: 10.1542/peds.2013-2000. Epub 2013 Nov 18. PMID 24249819
- [Background] Smulders CA, van Gestel JP, Bos AP. Are central line bundles and ventilator bundles effective in critically ill neonates and children? Intensive Care Med. 2013 Aug;39(8):1352-8. doi: 10.1007/s00134-013-2927-7. Epub 2013 Apr 25. PMID 23615702
- [Background] Schulman J, Stricof R, Stevens TP, Horgan M, Gase K, Holzman IR, Koppel RI, Nafday S, Gibbs K, Angert R, Simmonds A, Furdon SA, Saiman L; New York State Regional Perinatal Care Centers. Statewide NICU central-line-associated bloodstream infection rates decline after bundles and checklists. Pediatrics. 2011 Mar;127(3):436-44. doi: 10.1542/peds.2010-2873. Epub 2011 Feb 21. PMID 21339265
- [Background] Casanova D, Bardot J, Magalon G. Emergency treatment of accidental infusion leakage in the newborn: report of 14 cases. Br J Plast Surg. 2001 Jul;54(5):396-9. doi: 10.1054/bjps.2001.3593. PMID 11428769
- [Background] Collins CL, Barfield C, Horne RS, Davis PG. A comparison of nasal trauma in preterm infants extubated to either heated humidified high-flow nasal cannulae or nasal continuous positive airway pressure. Eur J Pediatr. 2014 Feb;173(2):181-6. doi: 10.1007/s00431-013-2139-8. Epub 2013 Aug 18. PMID 23955516
- [Background] Farquhar C, Armstrong S, Kim B, Masson V, Sadler L. Under-reporting of maternal and perinatal adverse events in New Zealand. BMJ Open. 2015 Jul 23;5(7):e007970. doi: 10.1136/bmjopen-2015-007970. PMID 26204910
- [Background] Raju TN, Suresh G, Higgins RD. Patient safety in the context of neonatal intensive care: research and educational opportunities. Pediatr Res. 2011 Jul;70(1):109-15. doi: 10.1203/PDR.0b013e3182182853. PMID 21386749
- [Background] Garland JS, Alex CP, Uhing MR, Peterside IE, Rentz A, Harris MC. Pilot trial to compare tolerance of chlorhexidine gluconate to povidone-iodine antisepsis for central venous catheter placement in neonates. J Perinatol. 2009 Dec;29(12):808-13. doi: 10.1038/jp.2009.161. Epub 2009 Oct 8. PMID 19812587
- [Derived] Yager H, Tauzin M, Durrmeyer X, Todorova D, Storme L, Debillon T, Casagrande F, Jung C, Audureau E, Layese R, Caeymaex L; SEPREVEN Study Group. Respiratory outcomes and survival after unplanned extubation in the NICU: a prospective cohort study from the SEPREVEN trial. Arch Dis Child Fetal Neonatal Ed. 2024 Oct 18;109(6):586-593. doi: 10.1136/archdischild-2023-326679. PMID 38636983
- [Derived] Jaloustre M, Cohen R, Biran V, Decobert F, Layese R, Audureau E, Le Sache N, Chevallier M, Boukhris MR, Bolot P, Caeymaex L, Tauzin M; with the SEPREVEN study Group. Determinants of morbidity and mortality related to health care-associated primary bloodstream infections in neonatal intensive care units: a prospective cohort study from the SEPREVEN trial. Front Pediatr. 2023 May 31;11:1170863. doi: 10.3389/fped.2023.1170863. eCollection 2023. PMID 37325351
- [Derived] Passini L, Le Bouedec S, Dassieu G, Reynaud A, Jung C, Keller ML, Lefebvre A, Katty T, Baleyte JM, Layese R, Audureau E, Caeymaex L; SEPREVEN Study Group. Error disclosure in neonatal intensive care: a multicentre, prospective, observational study. BMJ Qual Saf. 2023 Oct;32(10):589-599. doi: 10.1136/bmjqs-2022-015247. Epub 2023 Mar 14. PMID 36918264
- [Derived] Caeymaex L, Astruc D, Biran V, Marcus L, Flamein F, Le Bouedec S, Guillois B, Remichi R, Harbi F, Durrmeyer X, Casagrande F, Le Sache N, Todorova D, Bilal A, Olivier D, Reynaud A, Jacquin C, Roze JC, Layese R, Danan C, Jung C, Decobert F, Audureau E. An educational programme in neonatal intensive care units (SEPREVEN): a stepped-wedge, cluster-randomised controlled trial. Lancet. 2022 Jan 22;399(10322):384-392. doi: 10.1016/S0140-6736(21)01899-7. PMID 35065786
- [Derived] Caeymaex L, Lebeaux C, Roze JC, Danan C, Reynaud A, Jung C, Audureau E. Study on preventing adverse events in neonates (SEPREVEN): A stepped-wedge randomised controlled trial to reduce adverse event rates in the NICU. Medicine (Baltimore). 2020 Jul 31;99(31):e20912. doi: 10.1097/MD.0000000000020912. PMID 32756081